CLINICAL TRIAL: NCT03770455
Title: PDL-1 Inhibition With Avelumab and Concurrent Second-generation ADT in African Americans With Castrate-resistant Metastatic Prostate Cancer
Brief Title: Avelumab Plus 2nd-generation ADT in African American Subjects With mCRPC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early signs of progression and learned experience that the assumed time period between psa progression and radiographic progression was shorter than expected
Sponsor: Jodi Layton, MD (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor-Investigator, Jodi Layton, MD, Assistant Professor of Medicine, Tulane University School of Medicine
Organization: Tulane University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1236
Record Dates: First submitted 2018-10-05; First posted 2018-12-10 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — avelumab; abiraterone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab + 2nd generation ADT (Experimental): Avelumab 10mg/kg every 2 weeks (Q2W) + 2nd generation ADT
  Interventions: Drug: Avelumab; Drug: 2nd generation ADT (abiraterone or enzalutamide)

INTERVENTIONS:
Drug: Avelumab — Avelumab 10mg/kg every 2 weeks (Q2W) + 2nd generation ADT
  Other Names: Bavencio
Drug: 2nd generation ADT (abiraterone or enzalutamide) — 2nd generation ADT (abiraterone or enzalutamide)

SUMMARY:
This is a nonrandomized, open-label trial of avelumab in subjects with metastatic castration-resistant prostate cancer (mCRPC) experiencing PSA or radiographic progression while receiving 2nd generation ADT (abiraterone / enzalutamide/ apalutamide or darolutamide). Metastases must be radiographically evident by whole body bone scintigraphy or CT/MRI scan.

Thirteen African American subjects will be enrolled into the initial cohort.

If at least one positive response (PSA decrease by >50% and or radiographic per RECIST 1.1) is found, the study will be expanded to accrue a total of 27 patients. The trial will be conducted in accordance with Good Clinical Practices.

Subjects enrolled in the study will receive avelumab 10 mg/kg every 2 weeks (Q2W) and continue their previously started 2nd generation ADT (abiraterone or enzalutamide).

Treatment with avelumab will continue until documented confirmed disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, Investigator's decision to withdraw the subject, subject discontinuation from the study, noncompliance with trial treatment or procedure requirements, subject receives 52 administrations of avelumab (approximately 2 years), or administrative reasons requiring the cessation of treatment.

After the end of treatment, each subject will be followed for 30 days for AE monitoring (serious AEs will be collected for 90 days after the end of treatment or 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier). Subjects who discontinue treatment for reasons other than disease progression will remain on study and continue to undergo study-related disease assessments until documented disease progression, initiation of a new non-study prostate cancer treatment, withdrawal of consent, or becoming lost to follow-up. All subjects will enter survival follow up, and will be contacted at their regularly scheduled clinic visit, or by telephone approximately every 6 months, until death or withdrawal of consent or end of study.

DETAILED DESCRIPTION:
This is a nonrandomized, open-label trial of avelumab in subjects with metastatic castration-resistant prostate cancer (mCRPC) experiencing PSA or radiographic progression while receiving 2nd generation ADT (abiraterone / enzalutamide/ apalutamide or darolutamide). Metastases must be radiographically evident by whole body bone scintigraphy or CT/MRI scan.

Thirteen African American subjects will be enrolled into the initial cohort. If at least one positive response (PSA decrease by >50% and or radiographic per RECIST 1.1) is found, the study will be expanded to accrue a total of 27 patients. The trial will be conducted in accordance with Good Clinical Practices.

Subjects enrolled in the study will receive avelumab 10 mg/kg every 2 weeks (Q2W) and continue their previously started 2nd generation ADT (abiraterone or enzalutamide).

All subjects will undergo radiographic imaging assessments and PSA assessments to evaluate response to treatment at regular intervals. On study imaging will be assessed every 12 weeks. Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 will be adapted per the consensus guidelines of the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) as described in Appendix A/B to account for the tumor progression patterns seen in bone metastases in prostate cancer. PSA will be obtained every 2 weeks with PSA progression assessed per PCWG3.

Adverse events (AEs) will be monitored throughout the trial and graded in severity according to the guidelines outlined in the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

Treatment with avelumab will continue until documented confirmed disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, Investigator's decision to withdraw the subject, subject discontinuation from the study, noncompliance with trial treatment or procedure requirements, subject receives 52 administrations of avelumab (approximately 2 years), or administrative reasons requiring the cessation of treatment.

After the end of treatment, each subject will be followed for 30 days for AE monitoring (serious AEs will be collected for 90 days after the end of treatment or 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier). Subjects who discontinue treatment for reasons other than disease progression will remain on study and continue to undergo study-related disease assessments until documented disease progression, initiation of a new non-study prostate cancer treatment, withdrawal of consent, or becoming lost to follow-up. All subjects will enter survival follow up, and will be contacted at their regularly scheduled clinic visit, or by telephone approximately every 6 months, until death or withdrawal of consent or end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Must be of African descent; Black or African American: A person having origins in any of the black racial groups of Africa. Terms such as "Haitian" or "Negro" can be used in addition to "Black or African American."
2. Be willing and able to provide written informed consent for the trial.
3. Be ≥18 years of age on day of signing informed consent.
4. Have histologically or cytologically confirmed adenocarcinoma of the prostate without small cell histology. Diagnosis must be stated in a pathology report.
5. Have evidence of metastatic disease as determined by CT/MRI scans and/or bone metastases by whole body bone scintigraphy. (Use MRI if CT is contraindicated, and for imaging of the brain if clinically indicated).
6. Have documented disease progression within 3 months of screening, as determined by the Investigator, by means of at least one of the following:

   PSA progression as defined by a minimum of two rising PSA levels with an interval of ≥ 1 week between each assessment where the PSA value at screening should be ≥ 2 ng/mL.

   Radiographic disease progression in soft tissue or bone with or without PSA progression as determined by Recist 1.1 and/or PCWG3
7. Have ongoing androgen deprivation with serum testosterone < 50 ng/dL (< 2.0 nM). If the subject is currently being treated with Luteinising Hormone Releasing Hormone (LHRH) agonists or antagonists (for subjects who have not undergone an orchiectomy). This treatment must be continued throughout the study.
8. Be receiving and tolerating either abiraterone acetate, enzalutamide, apalutamide or darolutamide for at least 8 weeks prior to documented disease progression. Note: the 2nd generation ADT that the patient is currently progression on needs to be the first 2nd gen ADT used in the CRPC setting
9. Have a performance status of 0, 1 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale (Appendix D).
10. Male subjects of reproductive potential must agree practice abstinence from heterosexual activity OR use a highly effective method of contraception, starting at the time of informed consent and continue through 60 days after the last dose of study therapy (see section 6.1.1.)
11. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

Exclusion Criteria:

1. Is currently participating and receiving study therapy in a clinical trial, or has participated in a study of an investigational agent (and received study therapy or used an investigation device) within 4 weeks of the first dose of study treatment.
2. No more than one line of a 2nd generation ADT (abiraterone acetate /enzalutamide/ apalutamide/darolutamide) for mCRPC is permitted for study entry.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.

   Note: the following are allowed: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intraarticular injection); b. systemic corticosteroids at physiological doses < 10mg/day of prednisone or equivalent; c. steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
4. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to the first dose of trial treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to mAbs administered more than 4 weeks earlier.
5. Has had >2 prior systemic chemotherapy agents for mCRPC Note: chemotherapy in the metastatic hormone sensitive prostate cancer (mHSPC) setting is allowed
6. Prior surgery within 4 weeks of initiating study treatment Note: If subjects received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to the first dose of trial treatment.
7. Has any additional malignancy that has required active treatment in the last 3 years.

   Exceptions include: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or low-grade Ta or T1 urothelial carcinoma of that bladder that has undergone potentially curative therapy.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

   Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has an active autoimmune disease that might deteriorate when receiving an immune-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
10. Has had prior organ transplantation including allogenic stem-cell transplantation.
11. Has an active infection requiring systemic therapy.
12. Has active, clinically significant Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Patients with well controlled HIV will be allowed to be enrolled into the study.
13. Has Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test is positive).
14. Has received a live vaccine within 4 weeks of first dose of avelumab; live vaccines are prohibited throughout course of the trial. Inactivated vaccines are allowed.
15. Has known prior severe hypersensitivity to investigational product or component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.3 Grade > 3).
16. Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6months prior to enrollment), myocardial infarction (< 6months prior to enrollment), unstable angina, congestive heart failure (> New York Heart Association Classification Class II), or serious cardiac ventricular arrhythmia requiring medication.
17. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.3 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
18. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male based on biological distinctions not self-representation. Subject must have prostate cancer
Enrollment: 8 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jodi L Layton, MD, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane University School of Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: 2022
Access Criteria: To be determined pending publication

REFERENCES:
- [Background] Graff JN, Alumkal JJ, Drake CG, Thomas GV, Redmond WL, Farhad M, Cetnar JP, Ey FS, Bergan RC, Slottke R, Beer TM. Early evidence of anti-PD-1 activity in enzalutamide-resistant prostate cancer. Oncotarget. 2016 Aug 16;7(33):52810-52817. doi: 10.18632/oncotarget.10547. PMID 27429197
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Dominguez-Valentin M, Joost P, Therkildsen C, Jonsson M, Rambech E, Nilbert M. Frequent mismatch-repair defects link prostate cancer to Lynch syndrome. BMC Urol. 2016 Mar 24;16:15. doi: 10.1186/s12894-016-0130-1. PMID 27013479
- [Background] Raymond VM, Mukherjee B, Wang F, Huang SC, Stoffel EM, Kastrinos F, Syngal S, Cooney KA, Gruber SB. Elevated risk of prostate cancer among men with Lynch syndrome. J Clin Oncol. 2013 May 10;31(14):1713-8. doi: 10.1200/JCO.2012.44.1238. Epub 2013 Mar 25. PMID 23530095
- [Background] Pritchard CC, Mateo J, Walsh MF, De Sarkar N, Abida W, Beltran H, Garofalo A, Gulati R, Carreira S, Eeles R, Elemento O, Rubin MA, Robinson D, Lonigro R, Hussain M, Chinnaiyan A, Vinson J, Filipenko J, Garraway L, Taplin ME, AlDubayan S, Han GC, Beightol M, Morrissey C, Nghiem B, Cheng HH, Montgomery B, Walsh T, Casadei S, Berger M, Zhang L, Zehir A, Vijai J, Scher HI, Sawyers C, Schultz N, Kantoff PW, Solit D, Robson M, Van Allen EM, Offit K, de Bono J, Nelson PS. Inherited DNA-Repair Gene Mutations in Men with Metastatic Prostate Cancer. N Engl J Med. 2016 Aug 4;375(5):443-53. doi: 10.1056/NEJMoa1603144. Epub 2016 Jul 6. PMID 27433846
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Pritchard CC, Morrissey C, Kumar A, Zhang X, Smith C, Coleman I, Salipante SJ, Milbank J, Yu M, Grady WM, Tait JF, Corey E, Vessella RL, Walsh T, Shendure J, Nelson PS. Complex MSH2 and MSH6 mutations in hypermutated microsatellite unstable advanced prostate cancer. Nat Commun. 2014 Sep 25;5:4988. doi: 10.1038/ncomms5988. PMID 25255306
- [Background] Escudier B, Motzer RJ, Sharma P, Wagstaff J, Plimack ER, Hammers HJ, Donskov F, Gurney H, Sosman JA, Zalewski PG, Harmenberg U, McDermott DF, Choueiri TK, Richardet M, Tomita Y, Ravaud A, Doan J, Zhao H, Hardy H, George S. Treatment Beyond Progression in Patients with Advanced Renal Cell Carcinoma Treated with Nivolumab in CheckMate 025. Eur Urol. 2017 Sep;72(3):368-376. doi: 10.1016/j.eururo.2017.03.037. Epub 2017 Apr 12. PMID 28410865
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579
- [Background] Sartor et al. Overall Survival Analysis of African American and Caucasian Patients Receiving Sipuleucel-T: Preliminary Data from the Proceed Registry. J Urol, Vol 197: 4, April 2017.
- [Derived] Hawkins CM, Barata PC, Cotogno P, Davis G, Jaeger E, Ledet E, Miller P, Lewis B, Sartor O, Layton J. Black Patients with Metastatic Castrate-Resistant Prostate Cancer Have a Shorter Time Interval Between PSA and Clinical Progression on Novel Hormonal Therapies plus Avelumab. Oncologist. 2023 Mar 17;28(3):276-e158. doi: 10.1093/oncolo/oyac203. PMID 36210487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 25, 2019 - 11 September 2020
  Location: Tulane Cancer Center
Period: Overall Study
Arm/Group | Avelumab + 2nd Generation ADT
Started | 8
Completed | 5
Not Completed | 3
Not completed — Screen failures | 3

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab + 2nd Generation ADT
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Prostate-Specific Antigen (PSA) Response Greater Than or Equal to 50%
Description: The primary endpoint is a PSA response at 8 weeks or greater from starting study treatment and with a minimum of 3 treatments administered.
  A PSA response is defined as a ≥50% PSA decline at 8 weeks or greater from the time of starting study treatment. The two-stage minimax design of the study will be utilized to determine whether further investigation of the study drug is warranted.
Time Frame: 8 Weeks, 6 months
Population: Study closed early due to safety concerns. None of the participants reached the 8 weeks time point pre-specified for this analysis and hence PSA response data were not collected.
Arm/Group | Avelumab + 2nd Generation ADT
Number analyzed (Participants) | 0

2. Secondary Outcome: PSA Progression-free Survival (PFS)
Description: PSA progression-free survival (pPFS) defined as the time from enrollment until PSA progression by Prostate Cancer Working Group 3 (PCWG3) or death, whichever occurs earlier. Subjects without pPFS at the time of data cut-off will be censored at the date of last adequate cancer assessment. PSA progression-free survival will be reported using Kaplan-Meier estimates, with 95% confidence interval for median time-to-event.
Time Frame: pPFS will be assessed 12 months after enrollment of last subject.
Population: Study closed early due to safety concerns. Statistically underpowered and did not meet timeframe of pPFS assessed at 12 months after enrollment of last subject, so the investigators were not able to calculate PSA Progression-free Survival due to early closure, and none of the 5 participants had data to be summarized.
Arm/Group | Avelumab + 2nd Generation ADT
Number analyzed (Participants) | 0

3. Secondary Outcome: Radiographic Progression-free Survival (PFS)
Description: Radiographic progression-free survival (rPFS) defined as the time from enrollment until radiographic progression by PCWG3 or death, whichever occurs earlier. Subjects without rPFS at the time of data cut-off will be censored at the date of last known to be alive. Radiographic progression-free survival will be reported using Kaplan-Meier estimates, with 95% confidence interval for median time-to-event.
Time Frame: rPFS will be assessed 12 months after enrollment of last subject.
Population: Study closed early due to safety concerns. Statistically underpowered and did not meet timeframe of rPFS assessed at 12 months after enrollment of last subject, so the investigators were not able to calculate Radiographic Progression-free Survival due to early closure, and none of the 5 participants had data to be summarized.
Arm/Group | Avelumab + 2nd Generation ADT
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) defined as the time from enrollment until death on study. Subjects who are alive at the time of data cut-off will be censored at the date of last known to be alive. OS will be reported using Kaplan-Meier estimates, with 95% CI for median time-to-event.
Time Frame: Overall survival with be assessed at 3 years from time of enrollment of last study subject.
Population: Study closed early due to safety concerns. Statistically underpowered and did not meet timeframe of overall survival assessed at 3 years from time of enrollment of last study subject, so the investigators were not able to calculate Overall Survival due to early closure, and none of the 5 participants had data to be summarized.
Arm/Group | Avelumab + 2nd Generation ADT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | Avelumab + 2nd Generation ADT
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab + 2nd Generation ADT (N=5)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
L2 compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Severe pain from back to leg/sciatica (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab + 2nd Generation ADT (N=5)
Constipation (Gastrointestinal disorders) | 3 (6)
Fatigue (General disorders) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 3 (10)
Cramps (Musculoskeletal and connective tissue disorders) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin on feet (Skin and subcutaneous tissue disorders) | 1 (1)
Intermittent diarrhea (Gastrointestinal disorders) | 1 (1)
Localized rash bilateral elbows (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Hyperglycemia (General disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypokaelmia (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study did not reach target number of participants needed to reach target power for statistically reliable results due to poor recruitment during Coronavirus Disease 2019 (COVID-19) pandemic and early termination of study.

Study closed early due to safety concerns regarding rapid clinical progression of several participants, therefore, the secondary outcome measures were not analyzed and no data was reported for those outcome measures, so they were deleted from the study record.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03770455/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT03770455/ICF_001.pdf